CLINICAL TRIAL: NCT00586976
Title: A Phase II/III Study of Continuous Local Anesthetic Infusion in Median Sternotomy Following Cardiac Surgery
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Stopped by DSMB due to increased wound infection rate.
Sponsor: Mayo Clinic (Other)
Collaborators: Stryker Nordic (Industry)
Responsible Party: Gregory A. Nuttall, Mayo Clinic College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1107-05; Contract number 1a5777
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Cardiac Surgery
Keywords: pain, ropivacaine, infusion, sternotomy
MeSH Terms: conditions — Pain | interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Ropivicaine infusion into the sternal wound
  Interventions: Drug: Ropivacaine
- 2 (Placebo Comparator): Normal saline infusion into the sternal wound
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ropivacaine — 0.3% ropivacaine infusion at 4 ml/hr for 64 hours.
  Arms: 1
Drug: Normal saline — Normal saline infusion at 4 ml/hour for 64 hours.
  Arms: 2

SUMMARY:
Cardiac surgery is associated with pain in the post-operative period. We plan to conduct a study of local anesthetic, ropivacaine, infusion into the sternal wound in adult patients undergoing cardiac surgery to see if it will be safe and result in improved pain control and reduced time to extubation, duration of ICU and hospital stay.

DETAILED DESCRIPTION:
Background:

Cardiac surgery is associated with pain in the post-operative period. Recently the ability to infuse local anesthetic drugs into the area of the sternal wound has become available. The studies that have been done thus far have shown efficacy in controlling pain but have been too small to show clinically significant patient outcome differences.

Specific Aim:

We plan to conduct a phase II/III study of local anesthetic infusion into the sternal wound in adult patients undergoing cardiac surgery.

In the Phase II study, 40 patients will be enrolled in a prospective observational open label, dose escalation study of safety and efficacy of local anesthetic infusion into the sternal wound. Outcome measures for efficacy will be visual analog pain (VAP) scores and opioid consumption. Outcome measures for safety will be plasma ropivacaine concentrations and adverse events.

The dose determined in the phase II study will be used in the Phase III study. In this study, 200 patients will be enrolled in a double blind prospective, randomized, double blind; placebo controlled trial of local anesthetic infusion into the sternal wound. Outcome measures for efficacy will be visual analog pain (VAP) scores, opioid consumption, time to extubation, pulmonary function tests, duration of ICU and hospital stay, all cause morbidity and mortality. Outcome measure for safety will be adverse events.

Hypothesis:

Local anesthetic infusion into the sternal wound will be safe and result in improved pain control and reduced time to extubation, duration of ICU and hospital stay.

Significance:

This will be the first large randomized controlled clinical trial assessing outcomes with the use of local anesthetic infusion into the sternal wound in patients undergoing open-heart surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Be greater than 18 years of age
2. Be undergoing a cardiac surgical procedure via median sternotomy (i.e., exclude the occasional thoracotomy, since much greater pain with that surgical approach post-operatively)

Exclusion Criteria:

1. Are unable to grant informed consent or comply with study procedure
2. Are undergoing emergency open heart-surgery
3. Allergic to any of the excipients in ropivacaine, propofol, and fentanyl
4. Age < 18 years of age (children have dosing and toxicity concerns)
5. Are pregnant (pregnancy changes pain thresholds)
6. Taking preoperative opioids. (Opioid tolerant patients will require significantly more post-operative opioid use.)
7. Cirrhosis or hepatic failure (may have accumulation of local anesthetic in plasma due to decreased metabolism)
8. Patient receiving lidocaine infusion prior to surgery. (An extremely rare event)
9. Patients having a planned circulatory arrest for their surgical procedure (increased duration of intubation possible)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2005-07; Primary Completion 2007-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Visual analog pain | 64 hours

SECONDARY OUTCOMES:
drug toxicity | 64 hours
infection | 64 hours
narcotic usage | 64 hours

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A. Nuttall, M.D., Principal Investigator — Mayo Clinic College of Medicine
Locations (1):
- Mayo Clinic College of Medicine, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Agarwal S, Nuttall GA, Johnson ME, Hanson AC, Oliver WC Jr. A prospective, randomized, blinded study of continuous ropivacaine infusion in the median sternotomy incision following cardiac surgery. Reg Anesth Pain Med. 2013 Mar-Apr;38(2):145-50. doi: 10.1097/AAP.0b013e318281a348. PMID 23386053